CLINICAL TRIAL: NCT06682858
Title: Developing a Mechanistically Informed Therapy for Aversive Sensory Experiences with Autistic Youth
Brief Title: Developing a Novel Therapy for Aversive Sensory Experiences in Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 346716
Record Dates: First submitted 2024-10-25; First posted 2024-11-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Autism; Autism in Children
Keywords: sensory processing; anxiety; cognitive behavioural therapy; perception; autism
MeSH Terms: conditions — Autistic Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group Cognitive Behavioural Therapy (Experimental)
  Interventions: Behavioral: Group Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Group Cognitive Behavioural Therapy — Participants will complete 8 group sessions of a CBT-based intervention designed to help self-regulate sensory difficulties in autistic young people

SUMMARY:
The goal of this study is to assess whether a new psychological treatment can lead to changes in sensory experiences in autistic young people. Participants will complete a group intervention designed to help manage sensory difficulties and associated anxiety. Participants will also complete tasks before and after the intervention to assess whether the treatment can lead to changes in brain and behavioural responses to sensory experiences.

The main questions the study aims to answer are:

1. Does the intervention improve sensory difficulties and associated anxiety in autistic young people?
2. Does the intervention change brain and biological responses to sensory experiences in autistic young people?

Researchers will also collect feedback from participants to help improve the design and delivery of the treatment in future studies.

DETAILED DESCRIPTION:
The purpose of this study is to pilot a group-based cognitive behavioural therapy (CBT) intervention focused on managing sensory differences associated with autism. Another aim of this study is to test whether the intervention can modulate perceptual and neurophysiological markers (e.g. via electrocephalogram [EEG], heart rate and skin conductance) of sensory processing in autistic children and adolescents. A final aim will be to collect qualitative feedback from autistic young people with the aim of refining and improving the intervention for larger studies in the future.

The main aims of the study are:

1. To assess the feasibility of a novel CBT intervention for the management of sensory difficulties and associated anxiety in autistic youth.
2. To gather proof-of-concept data that the intervention can be used to modulate sensory neurophysiological and perceptual markers.
3. To gather qualitative feedback and PPIE to inform refinements on the design and delivery of the intervention for further studies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of autism
* Verbal/intellectual ability in average range
* Sufficient spoken English to be able to access the intervention
* Under the care of a local mental health service
* Not currently taking part in another psychological intervention

Exclusion Criteria:

* Verbal/intellectual ability below the average range
* Insufficient spoken English to be able to access the intervention
* Currently receiving a psychological intervention
* Individuals at high risk of harm to themselves or others

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Acceptability of the intervention will be assessed through study completion, an average of 1 year
  As this is a feasibility study, the primary outcome of interest is the acceptability of the intervention which will be assessed via drop-out rate and qualitative feedback

SECONDARY OUTCOMES:
Adolescent/Adult Sensory Profile (AASP) | Data collected on 2 visit days for each participant, before and after the intervention, about 12 weeks apart
  The Adolescent/Adult Sensory Profile (AASP) is a 60-item self-report questionnaire on sensory preferences and responses to sensory experiences. The AASP yields 4 subscale scores for sensory avoiding, sensitivity, seeking, and low registration. Raw total scores can range 60-300, with higher scores indicating greater sensory difficulties.
Revised Child Anxiety and Depression Scale (RCADS) | Data collected on 2 visit days for each participant, before and after the intervention, about 12 weeks apart
  The Revised Child Anxiety and Depression Scale (RCADS) is a 47-item youth self-report measure for anxiety and depression. Raw total scores can range 0-141, with higher scores indicating greater anxiety and/or depression. The RCADS can also yield subscales for separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder).
Interoception Sensory Questionnaire (ISQ-8) | Data collected on 2 visit days for each participant, before and after the intervention, about 12 weeks apart
  The Interoception Sensory Questionnaire short-form (ISQ-8) is an 8-item self-report questionnaire that measures interoceptive challenges (confusion about bodily states) in autistic individuals. Raw total scores can range 8-40 (T-score range 33-78), with higher scores indicating a greater difficulty with registering or interpreting interoceptive sensations.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edgington L, Hill V, Pellicano E. The design and implementation of a CBT-based intervention for sensory processing difficulties in adolescents on the autism spectrum. Res Dev Disabil. 2016 Dec;59:221-233. doi: 10.1016/j.ridd.2016.09.004. Epub 2016 Sep 14. PMID 27639063